CLINICAL TRIAL: NCT06028945
Title: Randomized Controlled Trial Evaluating the Impact of Virtual Reality Exposure Therapy on Epilepsy/Seizure-Specific Interictal Anxiety In People With Epilepsy
Brief Title: Evaluating the Impact of Virtual Reality Exposure Therapy on Epilepsy/Seizure-Specific Interictal Anxiety
Acronym: AnxEMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-5516
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy; Anxiety Disorders
Keywords: Epilepsy; Anxiety; Virtual Reality; Exposure Therapy; Cognitive Behavioural Therapy; Seizure; Interictal Anxiety
MeSH Terms: conditions — Epilepsy; Anxiety Disorders; Seizures

STUDY DESIGN:
Intervention Model Description: Interventional, Randomized, Pilot, Pragmatic, Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: VR-ET (Experimental): Group 1 will receive the VR-ET for up to 10 days while in the EMU and complete a set of questionnaires at the first visit and after the last day of VR. A researcher will conduct a short exit interview with participants about their experience during their second visit. There will be a one-month follow-up phone interview with a researcher and participants will complete a final set of questionnaires.
  Interventions: Device: HMD: Virtual Reality Exposure Therapy
- Group 2: Neutral Game (Active Comparator): Group 2 will have access to a VR device with a "neutral" game for up to 10 days while in the EMU and complete a set of questionnaires at the first visit and after the last day of VR. A researcher will conduct a short exit interview with participants about their experience during their second visit. There will be a one-month follow-up phone interview with a researcher and participants will complete a final set of questionnaires.
  Interventions: Device: HMD: Neutral Game

INTERVENTIONS:
Device: HMD: Virtual Reality Exposure Therapy — The virtual reality exposure therapy uses 360-degree videos delivered through a head mounted display (HMD). Participants will be matched with one of three available exposure hierarchies: Social Party Scenario, Subway Scenario, or Shopping Mall Scenario. Each hierarchy comprises seven 5-min scenes ordered in increasing intensity (from low to high anxiety). Participants are gradually exposed to scenes, viewed twice per day for up to 10 days, while rating their anxiety immediately before and after the exposures. Anxiety ratings will inform when participants may advance to the next level intensity in the exposure hierarchy.
  Arms: Group 1: VR-ET
Device: HMD: Neutral Game — The neutral game is a virtual-reality based game that is not designed to provoke anxiety. Participants assigned to the neutral game will play for 5 minutes twice per day for up to 10 days.
  Arms: Group 2: Neutral Game

SUMMARY:
The purpose of this randomized control trial is to evaluate the impact of Virtual Reality (VR) Exposure Therapy (ET) on people with epilepsy who experience epilepsy/seizure-specific (ES) interictal anxiety. The main questions it aims to answer are:

1. Can virtual reality exposure therapy (VR-ET) help reduce ES-interictal anxiety in this population?
2. Are the study procedures sufficiently simple for participants to follow?

Study Design Summary:

* Fourteen (14) participants will be randomized into either an Experimental arm (receiving VR-ET) or Control arm
* Participants will be expected to have VR-ET twice a day (5 min/session) for up to 10 days
* Participants will complete self-reported questionnaires about anxiety, depression, quality life, and avoidance behaviours at baseline (T0), after completing their VR program (T2), and at a one-month follow-up (T3).
* Participants will have a short interview with a researcher after completing their VR program (T2) as well as at a one-month follow-up (T3).

Researchers will attempt to answer the study questions based on outcome measures taken at various timepoints and qualitative feedback from interviews.

DETAILED DESCRIPTION:
BASELINE VISIT #1 (T0):

The first study visit will take place at the participant's bedside in the EMU with a member of the research team. The participant will be asked to complete several questionnaires including: demographic/health history, anxiety, depression, avoidance behaviours, and quality of life. The researcher will show the participant a short neutral video with the VR device and check for symptoms of motion sickness that might occur using a scale from 0 to 20. Next the participant will work with the researcher to identify the most appropriate exposure therapy scenario. Finally the participant will be randomized into either Group 1 (Experimental Group) or Group 2 (Control Group) and receive training on the VR system specific to their group assignment.

INTERVENTION (T1):

Participants will be encouraged to use the VR system throughout their EMU stay, twice per day for up to 10 days. Each session will involve using VR for approximately 5 minutes. The intervention may last fewer than 10 days if any participant is discharged early from the EMU, or (for Group 1 participants) all levels of the exposure therapy is completed in less than 10 days. Before and after each exposure, participants will be asked to rate their anxiety level on a scale from 0 to 100. After each exposure, participants will also be asked to rate any motion sickness that might result from using VR on a scale from 0 to 20.

POST-INTERVENTION VISIT #2 (T2)

The second study visit will take place after the participant's last VR session. Participants will be asked to repeat questionnaires from Visit #1 on anxiety, depression, avoidance behaviours, and quality of life. Participants will also complete questionnaires about sense of presence in VR and usability of the system. Finally participants will have a short interview with the researcher to discuss their experience using VR and any thoughts about whether the intervention had an impact on their anxiety.

1-MONTH FOLLOW-UP VISIT #3 (T3)

The third study visit will take place one (1) month after Visit #2. A researcher will follow-up with a phone interview and provide a link through email for participants to repeat baseline questionnaires about anxiety, depression, avoidance behaviours, and quality of life. However if participants prefer, they may request the researcher to record their responses to the questionnaires over the phone rather than completing the web-based questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are at least 18 years old
* Individuals admitted to the EMU
* Individuals who have self-reported anxiety related to having epilepsy or seizures
* Individuals who score <15 on the Fast Motion Sickness (FMS) after the VR neutral demo

Exclusion Criteria:

* Individuals with an unconfirmed epilepsy diagnosis
* Individuals with stereotaxic EEG monitoring
* Individuals with photosensitive epilepsy
* Individuals with open wounds on the face or cervical conditions or injuries that would make it unsafe for use the VR headset
* Individuals who have started an antidepressant, antianxiety drug, or medical marijuana in the last twelve weeks
* Individuals who cannot speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Fast Motion Sickness (FMS) Scale | Baseline (T0)
  A single assessment question where motion sickness (nausea and general discomfort) is rated on a visual analog scale ranging from 0 (no sickness at all) to 20 (severe sickness). This scale will be used as a measure of simulator sickness during baseline training.
Epilepsy Anxiety Survey Instrument (EASI) | Baseline (T0), Post-Intervention (T2), 1-Month Follow-Up (T3)
  An 18-item questionnaire designed specifically to assess anxiety in people with epilepsy. Scores can range from 0 to 54, where higher scores indicate more severe anxiety.
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) | Baseline (T0), Post-Intervention (T2), 1-Month Follow-Up (T3)
  A 6-item screening tool for major depressive disorder (MDD) in people with epilepsy. Scores can range from 6 to 24, where higher scores indicate more severe depression.
Liebowitz Social Anxiety Scale | Baseline (T0), Post-Intervention (T2), 1-Month Follow-Up (T3)
  A 24-item scale used to assess fear and avoidance of a range of social interactions and performance situations. Scores range from 0 to 144, where higher scores indicate more severe social anxiety.
GAD-7 | Baseline (T0), Post-Intervention (T2), 1-Month Follow-Up (T3)
  A 7-item scale used to screen for generalized anxiety disorder. Scores range from 0 to 21, where higher scores indicate more severe anxiety.
QOLIE - 31 | Baseline (T0), Post-Intervention (T2), 1-Month Follow-Up (T3)
  A 31-item questionnaire measuring overall quality of life including emotional well-being and role limitations in people with epilepsy. Scores range from 0 to 100, where higher scores reflect higher quality of life.
Mobility Inventory for Agoraphobia | Baseline (T0), Post-Intervention (T2), 1-Month Follow-Up (T3)
  On this instrument, 26 situations and locations (including shopping malls, public transit, and social gatherings) are rated for avoidance both when accompanied by a trusted companion and when alone. Average scores for each subscale (accompanied vs alone) range from 1 (never avoid) to 5 (always avoid). The instrument also collects information on panic attacks, with a score ranging from 1 (very mild) to 5 (extremely severe).
Subjective Units of Distress/Discomfort Scale (SUDS) | Intervention Period (T1)
  A single assessment question where level of anxiety is rated on a visual analog scale ranging from 0 (no distress; totally relaxed) to 100 (highest anxiety/distress that you have ever felt). This scale will be used to measure anxiety immediately before and after VR exposures.
Fast Motion Sickness (FMS) Scale | Intervention Period (T1)
  A single assessment question where motion sickness (nausea and general discomfort) is rated on a visual analog scale ranging from 0 (no sickness at all) to 20 (severe sickness). This scale will be used as a measure of simulator sickness immediately after using VR.
System Usability Scale (SUS) | Post-Intervention (T2)
  A 10-item survey that provides a quick assessment of the usability of various products and services, including hardware, software, mobile devices, websites and applications. Scores range from 0 to 100, with higher scores indicating higher level of usability.
Igroup Presence Questionnaire (IPQ) | Post-Intervention (T2)
  Several subscales to measure sense of presence, spatial presence, involvement, and experienced realism while in the virtual environment. Average scores for the different subscales range from 0 to 6, with higher scores indicating higher sense of presence/realism.
Post-Intervention Interview (approx. 15 min) | Post-Intervention (T2)
  The semi-structured exit interview will be conducted by a researcher the day after the participant has completed their final VR session. The purpose of this interview is to collect feedback on the VR-system usability and training, treatment delivery, overall experience, and (experimental arm only) effectiveness of VR exposure scenes. Participants will also be asked about the intervention's perceived change on their anxiety.
Follow-Up Interview (approx. 15 min) | 1-Month Follow-Up (T3)
  The follow-up phone interview will take place one month post-intervention. The researcher will call the participant and inquire about their general and ES-interictal anxiety levels, as well as their current levels of, and any perceived changes in, fear/comfort and avoidance of feared scenarios.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Bui, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Hingray C, McGonigal A, Kotwas I, Micoulaud-Franchi JA. The Relationship Between Epilepsy and Anxiety Disorders. Curr Psychiatry Rep. 2019 Apr 29;21(6):40. doi: 10.1007/s11920-019-1029-9. PMID 31037466
- [Result] Munger Clary HM. Anxiety and epilepsy: what neurologists and epileptologists should know. Curr Neurol Neurosci Rep. 2014 May;14(5):445. doi: 10.1007/s11910-014-0445-9. PMID 24652453
- [Result] Munger Clary HM, Giambarberi L, Floyd WN, Hamberger MJ. Afraid to go out: Poor quality of life with phobic anxiety in a large cross-sectional adult epilepsy center sample. Epilepsy Res. 2023 Feb;190:107092. doi: 10.1016/j.eplepsyres.2023.107092. Epub 2023 Jan 16. PMID 36701931
- [Result] Deng W, Hu D, Xu S, Liu X, Zhao J, Chen Q, Liu J, Zhang Z, Jiang W, Ma L, Hong X, Cheng S, Liu B, Li X. The efficacy of virtual reality exposure therapy for PTSD symptoms: A systematic review and meta-analysis. J Affect Disord. 2019 Oct 1;257:698-709. doi: 10.1016/j.jad.2019.07.086. Epub 2019 Jul 30. PMID 31382122
- [Result] Tychsen L, Thio LL. Concern of Photosensitive Seizures Evoked by 3D Video Displays or Virtual Reality Headsets in Children: Current Perspective. Eye Brain. 2020 Feb 11;12:45-48. doi: 10.2147/EB.S233195. eCollection 2020. PMID 32104130
- [Result] Gribkoff VK, Lum-Ragan JT. Evidence for nitric oxide synthase inhibitor-sensitive and insensitive hippocampal synaptic potentiation. J Neurophysiol. 1992 Aug;68(2):639-42. doi: 10.1152/jn.1992.68.2.639. PMID 1382122
- [Result] McConnell EA. Assessing a quadriplegic's severe headache. Nursing. 1990 Jan;20(1):84-7. No abstract available. PMID 2300295
- [Result] Gray HG, Tchao D, Lewis-Fung S, Pardini S, Harris LR, Appel L. Virtual Reality Therapy for People With Epilepsy and Related Anxiety: Protocol for a 3-Phase Pilot Clinical Trial. JMIR Res Protoc. 2023 Jan 24;12:e41523. doi: 10.2196/41523. PMID 36692939
- [Result] Tchao D, Lewis-Fung S, Gray H, Pardini S, Harris LR, Appel L. Describing epilepsy-related anxiety to inform the design of a virtual reality exposure therapy: Results from Phase 1 of the AnxEpiVR clinical trial. Epilepsy Behav Rep. 2023 Jan 16;21:100588. doi: 10.1016/j.ebr.2023.100588. eCollection 2023. PMID 36794093
- See also: EASI-18 — https://www.ilae.org/files/dmfile/EASI-18.pdf
- See also: Liebowitz Social Anxiety Scale — https://psychology-tools.com/test/liebowitz-social-anxiety-scale
- See also: Mobility Inventory for Agoraphobia — https://cpb-us-w2.wpmucdn.com/web.sas.upenn.edu/dist/6/184/files/2017/03/Mobility-Inventory-1zjichf.pdf
- See also: Subjective Units of Distress/Discomfort Scale (SUDS) — https://www.disordersofmood.com/pdf/SUDS.pdf
- See also: System Usability Scale (SUS) — https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html
- See also: Igroup Presence Questionnaire (IPQ) — http://www.igroup.org/pq/ipq/items.php
- See also: Fast Motion Sickness Scale (FMS) — https://pubmed.ncbi.nlm.nih.gov/21901938/
- See also: GAD-7 — https://adaa.org/sites/default/files/GAD-7_Anxiety-updated_0.pdf